CLINICAL TRIAL: NCT04029285
Title: The Effects of Exergaming on Pain, Postural Control, Technology Acceptance and Flow Experience in Older People With Chronic Musculoskeletal Pain: a Randomised Controlled Trial
Brief Title: Exergaming Experience of Older People With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Alasdair MacSween, Principal Lecturer (Research Governance), Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ExergamingOldPeople
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Pain Disorder
Keywords: Exergaming; Exercise Therapy; Musculoskeletal Pain; Aged, Aged 80 and Over; Postural Balance; Flow state experience; Technology acceptance; Heart Rate
MeSH Terms: conditions — Musculoskeletal Pain; Collagen Diseases | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the control group (TGB) or the experimental group (exergaming) in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Gym Based exercise - Control (Other): Twice weekly sessions of TGB exercise for six weeks.
  Interventions: Other: Exergaming
- Exergaming (Experimental): Twice weekly sessions of exergames for six weeks.
  Interventions: Other: Exergaming

INTERVENTIONS:
Other: Exergaming — The exergaming group played six IREX® exergames. Those in the TGB group performed exercises that were matched to the IREX® exergames for: movement patterns required, physiological demands, sequence, duration and mode of exercise by adopting open and closed kinetic chain movements, in the same range and loading, across both groups. Each IREX® exergame was played for two minutes and was repeated three times within a session. TGB exercise was conducted in sets of two minutes duration, repeated three times within a session. In both groups participants were given rest periods of 10 to 30 seconds, or longer, if required, between exergames or TGB exercise sets.

SUMMARY:
Chronic musculoskeletal pain is debilitating and can lower the quality of life in older people. Therapeutic benefits have been reported from exergaming used as an intervention for rehabilitation or alternative to exercise. This study investigated the effects of exergaming in comparison with those of standard exercise on pain, postural control, technology acceptance and flow experience in older people with musculoskeletal pain.

DETAILED DESCRIPTION:
Study design: A prospective, randomized, controlled two-arm trial design: Group 1) exergaming with the Interactive Rehabilitation and Exercise System (IREX®) and Group 2) traditional gym-based exercise (TGB).

Ethical Approval was sought from and granted by the School of Health and Social Care Research Governance and Ethics Committee at Teesside University on 20th September 2010 The study was conducted in the Physiotherapy Research Laboratory, Constantine Building, Teesside University.

Participants were recruited by non-direct contacts from nine local community groups in the Middlesbrough area.

Sixty-one potential participants were screened for eligibility. Four were excluded due to not meeting the eligibility criteria and three did not attend scheduled sessions. Fifty-four (42 females and 12 males, age: 71 ± 5 years) were allocated to either exergaming with the IREX™ (n = 27) or TGB (n = 27).

Procedure

On arrival for data collection at the Physiotherapy Research Laboratory at Teesside University, participants were asked if they had further questions about the study. These questions, if any, were answered. The study Consent Form was then signed. Participants' demographic details and all outcome measures were recorded, after which the participants were randomised by stratified blind-card allocation (picking a sealed opaque envelope).

Data extraction

Range and Standard Deviation (SD) of Centre of Pressure (CoP) displacements in the anterior-posterior (AP) and medio-lateral (ML) directions (CoPAP SD, CoPAP range, CoPML SD, CoPML range - all mm) and the resultant CoP velocity (mm.sec-1) were extracted from the force platform using Bioware software (Kistler™), after low-pass filtering of the raw data at 10 Hz. CoP velocity (mm.sec-1) was calculated.

Statistical analysis

Data was analysed with Version 19 of the Statistical Package for the Social Sciences (SPSS, Chicago, Illinois, USA). Analysis of covariance (ANCOVA) was used to assess between-group final scores for each outcome measure used with baseline scores as covariate. Variables that did not meet the assumption of homogeneity of variance were analysed by two-way independent measures ANOVA with blocking using mean splits of scored pre-measures. Mixed analysis of variance (ANOVA) was used to determine any within-subject changes over time. All analyses used a significance level of 0.05. The effect size measure epsilon squared was used, where values of 0.01, 0.06 and 0.14 were interpreted as small, moderate and large.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged 65 years or over
* able to walk unassisted (i.e. did not use, or require, any walking aids) for at least 0.5 of a mile
* having musculoskeletal pain in two or more joints, of more than 12 weeks duration

Exclusion Criteria:

* diagnosis (or suspicion) of any systemic conditions that may cause pain in two or more joints
* of more than 12 weeks duration (such as cancer, rheumatic or neurological disease or condition)
* self-report of current (or history) of any condition or injury which would contra- indicate participation in the exercises under study
* inability (or any doubt of ability) to give informed consent
* inability to read and write English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2011-09-16 (Actual)

PRIMARY OUTCOMES:
Change in score, on each cluster included in the Multi Affect and Pain Survey (MAPS) questionnaire (Clark, 2002). | Change in MAPS Cluster Score, from baseline to six weeks
  MAPS comprises three superclusters reflecting three major aspects of pain: somatosensory, emotional and well-being.
  1. somatosensory supercluster contains 17 clusters with 57 descriptors of painful sensory qualities
  2. emotional supercluster has 8 clusters with 26 descriptors of negative emotional qualities
  3. well-being supercluster has 5 clusters with 18 descriptors of positive affect, and health.
  Descriptors are presented as statements and participants rate how closely each comes to describing how they feel on a six point scale (from 0 (Not at all) to 5 (Very much so)). Descriptor scores are summed to give Cluster scores. An increased score in somatosensory and emotional clusters reflects a worsening, in well-being it reflects an improvement.
Change in Pain intensity (within previous 30 days) rating | Change in Pain intensity (within previous 30 days) rating, from baseline to six weeks
  Participants rated the intensity of their pain (within previous 30 days) on a 0-10 scale where 10 is the WORST POSSIBLE PAIN. An increased score represents greater pain.
Change in Pain intensity (at present time) rating | Change in Pain intensity (within previous 30 days) rating, from baseline to six weeks
  Participants rated the intensity of their pain (within previous 30 days) on a 0-10 scale where 10 is the WORST POSSIBLE PAIN. An increased score represents greater pain.
Change in rate of change of centre of pressure (mm.s-1) location - eyes open. | Change in centre of pressure velocity (mm.s-1) (eyes open), from baseline to six weeks
  Centre of pressure velocity (mm.s-1) is the rate at which the centre point of force (measured on a Kistler™ Force Plate) moves, as the participant stands on the force plate with their eyes open.
  It is quantified in mm.s-1 and an increase represents faster movements and hence more rapid corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in standard deviation of centre of pressure (mm) location measurements in the anterio-posterior direction - eyes open. | Change in standard deviation of centre of pressure (mm) location measurements in the anterio-posterior direction (eyes open), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes open. The location of the CoP changes in the anterio-posterior direction (forwards to backwards) if the person sways forward and backward. The variability in the magnitude of sway is reflected in the Standard Deviation of this measure.
  It is quantified in mm and an increased variation in movement means that more varied corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in range of centre of pressure (mm) location measurements in the anterior-posterior direction - eyes open. | Change in range of centre of pressure (mm) location measurements in the anterior-posterior direction (eyes open), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes open. The location of the CoP changes in the anterio-posterior direction (forwards to backwards) if the person sways forward and backward. The extent of maximal and minimal magnitude of sway is reflected in the Range of this measure.
  It is quantified in mm and an increase represents larger movements occurred and so correspondingly larger corrections of balance are required, to maintain equilibrium and hence postural control has worsened.
Change in standard deviation of centre of pressure (mm) location measurements in the medio-lateral direction - eyes open. | Change in standard deviation of centre of pressure (mm) location measurements in the medio-lateral direction (eyes open), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes open. The location of the CoP changes in the medio-lateral direction (side-to-side) if the person sways from side to side. The variability in the magnitude of sway is reflected in the Standard Deviation of this measure.
  It is quantified in mm and an increased variation in movement means that more varied corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in range of centre of pressure (mm) location measurements in the medio-lateral direction - eyes open. | Change in range of centre of pressure (mm) location measurements in the medio-lateral direction (eyes open), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes open. The location of the CoP changes in the medio-lateral direction (side-to-side) if the person sways from side to side. The extent of maximal and minimal magnitude of sway is reflected in the Range of this measure.
  It is quantified in mm and an increase represents larger movements occurred and so correspondingly larger corrections of balance are required, to maintain equilibrium and hence postural control has worsened.
Change in rate of change of centre of pressure (mm.s-1) location - eyes closed. | Change in rate of change of centre of pressure (mm.s-1) location (eyes closed), from baseline to six weeks
  Centre of pressure velocity (mm.s-1) is the rate at which the centre point of force (measured on a Kistler™ Force Plate) moves, as the participant stands on the force plate with their eyes closed.
  It is quantified in mm.s-1 and an increase represents faster movements and hence more rapid corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in standard deviation of centre of pressure (mm) location measurements in the anterio-posterior direction - eyes closed. | Change in standard deviation of centre of pressure (mm) location measurements in the anterio-posterior direction (eyes closed), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes closed. The location of the CoP changes in the anterio-posterior direction (forwards to backwards) if the person sways forward and backward. The variability in the magnitude of sway is reflected in the Standard Deviation of this measure.
  It is quantified in mm and an increased variation in movement means that more varied corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in range of centre of pressure (mm) location measurements in the anterior-posterior direction - eyes closed. | Change in range of centre of pressure (mm) location measurements in the anterior-posterior direction(eyes closed), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes closed. The location of the CoP changes in the anterio-posterior direction (forwards to backwards) if the person sways forward and backward. The extent of maximal and minimal magnitude of sway is reflected in the Range of this measure.
  It is quantified in mm and an increase represents larger movements occurred and so correspondingly larger corrections of balance are required, to maintain equilibrium and hence postural control has worsened.
Change in standard deviation of centre of pressure (mm) location measurements in the medio-lateral direction - eyes closed. | Change in standard deviation of centre of pressure (mm) location measurements in the medio-lateral direction (eyes closed), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes closed. The location of the CoP changes in the medio-lateral direction (side-to-side) if the person sways from side to side. The variability in the magnitude of sway is reflected in the Standard Deviation of this measure.
  It is quantified in mm and an increased variation in movement means that more varied corrections of balance are required to maintain equilibrium and hence postural control has worsened.
Change in range of centre of pressure (mm) location measurements in the medio-lateral direction - eyes closed. | Change in range of centre of pressure (mm) location measurements in the medio-lateral direction(eyes closed), from baseline to six weeks
  Centre of pressure (CoP) is the centre point of force (measured on a Kistler™ Force Plate) as the participant stands on the force plate with their eyes closed. The location of the CoP changes in the medio-lateral direction (side-to-side) if the person sways from side to side. The extent of maximal and minimal magnitude of sway is reflected in the Range of this measure.
  It is quantified in mm and an increase represents larger movements occurred and so correspondingly larger corrections of balance are required, to maintain equilibrium and hence postural control has worsened.
Change in score on each domain included in the Technology Acceptance: United Theory of Acceptance and Use of Technology (UTAUT) questionnaire (Venkatesh, 2003). | Change in score on each domain included in the Technology Acceptance: United Theory of Acceptance and Use of Technology (UTAUT) questionnaire, from baseline to six weeks
  The UTAUT comprises statements rated on a 7-point Likert scale, 1 strongly disagree to 7 strongly agree, grouped into six domains.
  1. performance expectancy, the belief that using a system will help improve performance,
  2. effort expectancy, how easy it is to use the technology
  3. social influence, how much the user believes others think they should use the technology
  4. facilitation conditions, how much the user believes they should use the technology,
  5. self-efficacy, how capable the user feel to use the technology
  6. behavioural intention, intention to use the technology again.
  Statement ratings are summed to give Domain scores. An increased score in any Domain reflects an increase in acceptance (positive outcome in respect of technology usage).
Change in score on each sub-scale included in the Flow State Scale (FSS) (Jackson and Marsh, 1996). | Change in score on each sub-scale included in the Flow State Scale questionnaire, from baseline to six weeks
  FSS comprises 36 questions rated on a 5-point Likert scale 1 strongly disagree to 5 strongly agree, grouped into nine subscales.
  1. autotelic experience, the intrinsically rewarding experience doing a task
  2. clear goals, clearly confident of action
  3. challenge-skill-balance, balance between skills and challenge
  4. concentration at task, complete control on performing a task
  5. control, at full focus at the task
  6. unambiguous feedback, feedback on performing a task
  7. action-awareness-merging, immediate, direct and clear observations whilst performing a task
  8. transformation of time, sense of time speeds or slows, becomes irrelevant or out of one's awareness
  9. loss of self consciousness, sense of not being concerned with oneself while engaged in a task
  Question ratings are summed to give subscale score. An increased score in any subscale reflects an increase in the experience of Flow State (a positive outcome in respect of experience of any activity).

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair MacSween, Principal Investigator — Teesside University
Locations (1):
- Teesside University, School of Health and Social Care, Middlesbrough, Cleveland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark CW, Yang JC, Tsui SL, Ng KF, Clark SB. Unidimensional pain rating scales: a multidimensional affect and pain survey (MAPS) analysis of what they really measure. Pain. 2002 Aug;98(3):241-247. doi: 10.1016/S0304-3959(01)00474-2. PMID 12127025
- [Background] Jackson SA. Toward a conceptual understanding of the flow experience in elite athletes. Res Q Exerc Sport. 1996 Mar;67(1):76-90. doi: 10.1080/02701367.1996.10607928. PMID 8735997
- [Background] Shamliyan TA, Wang SY, Olson-Kellogg B, Kane RL. Physical Therapy Interventions for Knee Pain Secondary to Osteoarthritis [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Nov. Report No.: 12(13)-EHC115-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK114568/ PMID 23213666
- [Derived] Ditchburn JL, van Schaik P, Dixon J, MacSween A, Martin D. The effects of exergaming on pain, postural control, technology acceptance and flow experience in older people with chronic musculoskeletal pain: a randomised controlled trial. BMC Sports Sci Med Rehabil. 2020 Oct 9;12:63. doi: 10.1186/s13102-020-00211-x. eCollection 2020. PMID 33062284